



### INFORMED CONSENT FORM

to Participate in Research, and

### **AUTHORIZATION**

to Collect, Use, and Disclose Protected Health Information (PHI)

| Introduction | |
|---|---|
| Name of person seeking your consent: | |
| Place of employment & position: | |
| GENERAL INFORMATION ABOUT THIS STUDY | |
| 1. Name of Participant ("Study Subject") | |
| 2. What is the title of this research study (this "Research Study")? | |
| The Effects of Intranasal Testosterone (Natesto™) for Treatment of Hypogonadism on Mai<br>Spermatogenesis | intenance of |
| 3. Whom do you call if you have questions about this Research Study (the "Stud | dy Team")? |
| Principal Investigator: Kevin Campbell | |
| 4. Who is naving for this Bosparch Study? | |

4. Who is paying for this Research Study?

The sponsor is the University of Florida.

#### 5. In general, what do you need to know about this Research Study?

Agreeing to become involved in any research is always voluntary. By signing this form, you are not waiving any of your legal rights. If you decide not to participate in this research, you will not be penalized in any way and you will not lose any benefits to which you are entitled. If you have questions about your rights as a research subject, please call the University of Florida Institutional Review Board (IRB) office at (352) 273-9600.

#### a) In general, what is the purpose of the research? How long will you be involved?

To determine if Natesto<sup>™</sup> can alleviate the symptoms of decreased energy, libido, decreased muscle mass, and lower bone mineral density, without affecting the ability to recover sperm production, in men who have stopped testosterone hormone therapy. Men will be started on stimulatory medical

IRB Project #:IRB202102979 

IRB Version: 08/13/2021 PI Version: 05/09/2022



therapy to induce recovery of sperm production, consistent with the standard of care. Natesto<sup>™</sup> has been shown to maintain sexual hormones at appropriate levels for sperm production without suppression in clinical trials. This medication will be offered in combination with the sperm stimulatory therapy to assist with hypogonadal symptoms while halting their routine form of testosterone.

### b) What is involved with your participation, and what are the procedures to be followed in the research?

Your participation will involve the standard of care for sperm stimulation following testosterone suppression. You will have routine hormone blood draws at 3 month intervals with semen analyses and symptom assessment through questionnaires. No procedures will be performed as a part of this study. You involvement with this study will involve you taking intranasal testosterone to combat your hypogonadal symptoms while on the standard of care medications to improve your sperm production.

#### c) What are the likely risks or discomforts to you?

Past studies have shown minor discomforts associated with Natesto<sup>TM</sup>. The most common adverse reaction includes elevated prostate specific antigens (PSA), headache, runny nose, nasal discomfort, or bleeding nasopharyngitis, upper respiratory tract infection, sinusitis, bronchitis, and nasal scab.

There are some risks associated with blood draws including pain, bruising, infection, lightheadedness, fainting, blood clots, and bleeding or other local site reactions.

The risk of stopping your current androgen replacement therapy (testosterone) includes low energy, low sex drive, and irritability.

#### d) What are the likely benefits to you or to others from the research?

The benefits of participating in this study may be: alleviation of hypogonadal symptoms associated with spermatogenesis stimulation. The hypogonadal symptoms include decreased energy, libido, muscle mass, and bone mineral density.

## e) What are the appropriate alternative procedures or courses of treatment, if any, that might be helpful to you?

The alternative procedures or treatments include the standard of care (high-dose HCG, anastrozole, and FSH or clomiphene) without intranasal testosterone.

# Additional and more detailed information is provided within the remainder of this Informed Consent form. Please read before deciding if you wish to participate in this study.

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

#### WHAT CAN YOU EXPECT IF YOU PARTICIPATE IN THIS STUDY?



# 6. What will be done as part of your normal clinical care (even if you did not participate in this Research Study)?

If you did not participate in this study and where to continue with normal clinical care, the clinical course would be identical except for the lack of intranasal testosterone and symptom assessment with questionnaires.

You would continue with clinic visits and undergo 3 month assessments including medical evaluations with a history and physical, hormone evaluation through bloodwork, and semen parameter evaluation with a semen analysis.

#### 7. What will be done only because you are in this Research Study?

Should you choose to be involved with this study, you will continue the standard of care with the addition of administering daily intranasal testosterone and completing symptom questionnaires every three months.

Participation in the study is completely voluntary. It will last approximately 26 weeks and consistent of clinic visits. The first clinic visit will consist of a medical evaluation performed by the UF Fertility team. At this time, blood will be drawn to measure testosterone levels, and other hormones. You will also be scheduled to perform a semen analysis shortly after the visit if you have not already had a recent test. During the course of the visit you will fill out 4 questionnaires – the IIEF, IPSS, ADAM, and SF36, They physician will go over in detail, that you must stop all testosterone and androgen therapy treatment for 4 weeks prior to initiating the study.

The next clinic visit will occur after 14 weeks (+/- 7 days). This visit will similarly include a medical evaluation, blood draw to evaluate hormones, and scheduling of an additional semen analysis. The questionnaires initially filled out will be updated.

The subsequent clinic visit will occur at 26 weeks (+/- 7 days). This visit will similarly include a medical evaluation, blood draw to evaluate hormones, and scheduling of an additional semen analysis. The questionnaires again will be updated.

Participants will be able to drop out of the study at any time should they desire or if they achieve a clinical pregnancy with their partner.

If any identifiable information is collected as part of this research, it is possible that your research information or specimens, with all personally identifiable information removed, could be used for future research studies or distributed to another investigator for future research studies without additional informed consent from you or your legally authorized representative.

If you have any questions now or at any time during this Research Study, please contact one of the Research Team members listed in question 3 of this form.

#### 8. What identifiable health information will be collected about you and how will it be used?

The Research Team will collect: demographic information, results of physical exams, hormone blood tests (FSH, LH, testosterone, estradiol, prolactin, CBC), semen analyses, and medical history.

The Research Team may collect this information from other healthcare providers, such as laboratories, which are a part of this research, as well as healthcare providers that are not part of this research (other

IRB Project #:IRB202102979 IRB Version: 08/13/2021

PI Version: 05/09/2022



doctors, hospitals or clinics). Other professionals at the University of Florida or Shands Hospital who provide study-related care, and the University of Florida Institutional Review Board (IRB), may also collect your health information.

The Research Team listed in question 3 above will use or share your health information as described below to carry out this research study.

#### 9. With whom will this health information be shared?

This health information may be shared with:

- the study sponsor (listed in Question 4 of this form);
- United States governmental agencies which are responsible for overseeing research, such as the Food and Drug Administration, the Department of Health and Human Services, and the Office of Human Research Protections;
- government agencies which are responsible for overseeing public health concerns, such as the Centers for Disease Control and federal, state and local health departments,
- Your insurance company for purposes of obtaining payment,
- the IRB that reviewed this Research Study and ensures your rights as a Study Subject are protected.

Otherwise, your identifiable health information will not be shared without your permission unless required by law or a court order. Once your health information is shared with those listed above, it is possible that they could share it without your permission because it would no longer be protected by the federal privacy law.

#### 10. How long will you be in this Research Study?

You will be in this research study for 26 weeks. You participation period may be shorter should you have a clinical pregnancy during that time or choose to withdraw from the study.

This Authorization to use and share your health information expires at the end of the study, unless you revoke it (take it back) sooner.

#### 11. How many people are expected to take part in this Research Study?

30 people are expected to take part in this Research Study.

# WHAT ARE THE RISKS AND BENEFITS OF THIS STUDY AND WHAT ARE YOUR OPTIONS?

#### 12. What are the possible discomforts and risks from taking part in this Research Study?

The risk in this study involve failure to relieve hypogonadal symptoms while on the medication.

Other possible risks to you may include: local adverse effects of intranasal testosterone as listed previously in this consent

The most common adverse reactions (incidence >3%) are: PSA increased, headache, rhinorrhea, epistaxis, nasal discomfort, nasopharyngitis, bronchitis, upper respiratory tract infection, sinusititis, and nasal scab.

IRB Project #:IRB202102979 

IRB Version: 08/13/2021 PI Version: 05/09/2022



This Research Study may also include risks that are unknown at this time.

Please note, participating in more than one research study or project may further increase the risks to you. If you are already enrolled in a research study, please inform one of the Research Team members listed in question 3 of this form or the person reviewing this consent with you before enrolling in this or any other research study or project.

During the study, the Research Team will notify you of new information that may become available and might affect your decision to remain in the study.

The University of Florida is required by law to protect your health information. Your health information will be stored in locked filing cabinets or on computer servers with secure passwords, or encrypted electronic storage devices, as required by University policy. However, there is a slight risk that information about you could be released inappropriately or accidentally. Depending on the type of information, a release could upset or embarrass you, or possibly affect your ability to get insurance or a job.

If you wish to discuss the information above or any discomforts you may experience, please ask questions now or call one of the Research Team members listed in question 3 in this form.

#### 13a. What are the potential benefits to you for taking part in this Research Study?

The benefits of participating in this study may be: alleviation of hypogonadal symptoms associated with spermatogenesis stimulation. The hypogonadal symptoms include decreased energy, libido, muscle mass, and bone mineral density.

#### 13b. How could others possibly benefit from this Research Study?

If NatestoTM demonstrates symptom relief of hypogonadism while patients are suspect their previous forms of testosterone in order to stimulate spermatogenesis, this may become a recommended treatment pathway for this population of men.

#### 13c. How could the Research Team members benefit from this Research Study?

In general, presenting research results helps the career of a researcher. Therefore, the Research Team listed in question 3 of this form may benefit if the results of this Research Study are presented at scientific meetings or in scientific journals.

The principal investigator has no conflict of interests in this study.

#### 14. What other choices do you have if you do not want to be in this study?

If you did not participate in this study and where to continue with normal clinical care, the clinical course would be identical except for the lack of intranasal testosterone and symptom assessment with questionnaires.

You would continue with clinic visits and undergo 3 month assessments including medical evaluations with a history and physical, hormone evaluation through bloodwork, and semen parameter evaluation with a semen analysis.

You may also refuse to authorize the use of your health information, but if you refuse, you may not be allowed to be in this research study or receive any research-related treatment that is only available in this



research study. However, your decision not to sign this Authorization will not affect any other treatment you may be eligible to receive.

#### 15a. Can you withdraw from this study?

You may withdraw your consent and stop participating in this Research Study at any time. If you do withdraw your consent, there will be no penalty to you, and you will not lose any benefits to which you are otherwise entitled. If you decide to withdraw your consent to participate in this Research Study for any reason, please contact the Research Team listed in question 3 of this form. They will tell you how to safely stop your participation.

You can also change your mind and take back this Authorization at any time by sending a written notice to the Research Team listed in question 3 of this form to let them know your decision. If you take back this Authorization, the Research Team may only use and disclose your health information already collected for this research study. No additional health information about you will be collected or disclosed to the Research Team. However, if you take back this Authorization, you may not be able to continue in this study. Please discuss this with a member of the Research Team listed in question #3.

#### 15b. Can the Principal Investigator withdraw you from this Research Study?

You may be withdrawn from this Research Study without your consent for the following reasons:

• Failure to obtain hormonal blood draws, semen analyses, or questionnaire completion.

#### WHAT ARE THE FINANCIAL ISSUES IF YOU PARTICIPATE?

#### 16. If you choose to take part in this Research Study, will it cost you anything?

The cost of participating in this study will be the cost of purchasing the Natesto<sup>™</sup> medication. A prescription will be ordered for you. Should your insurance not cover the medication or Natesto<sup>™</sup>, you will be responsible for the cost of the medication. The cost of Natesto<sup>™</sup> without insurance coverage is \$140 per month. This will cost \$840 for the entirety of the 6 month study if no financial assistance is provided.

There may be costs associated with the healthcare you receive while you are participating in this study. At least one of the protocol-required items, services or procedures that will generate charges at UF Health are considered to be conventional care that you would have received even if you chose not to participate in this study.

In addition, one or more protocol-required items, services or procedures will be provided by the sponsor at no charge to you.

If you receive any healthcare at UF Health that is not related to this study, this care will be billed as usual. If you feel you have received a bill related to this study in error, please contact the Principal Investigator.

#### 17. Will you be paid for taking part in this Research Study?

You will not be paid for taking part in this research study.

IRB Project #:IRB202102979 IRB Version: 08/13/2021 PI Version: 05/09/2022 



#### 18. What if you are injured while in this Research Study?

If you are injured as a direct result of your participation in this study, only the professional services that you receive from any University of Florida Health Science Center healthcare provider will be provided without charge. These healthcare providers include physicians, physician assistants, nurse practitioners, dentists or psychologists. Any other expenses, including Shands hospital expenses, will be billed to you or your insurance provider.

You will be responsible for any deductible, co-insurance, or co-payments. Some insurance companies may not cover costs associated with research studies or research-related injuries. Please contact your insurance company for additional information.

The Principal Investigator will determine whether your injury is related to your participation in this study.

No additional compensation is routinely offered. The Principal Investigator and others involved in this study may be University of Florida employees. As employees of the University, they are protected under state law, which limits financial recovery for negligence.

Please contact one of the research team members listed in question 3 of this form if you experience an injury or have questions about any discomforts that you experience while participating in this study.



### **SIGNATURES**

| As an investigator or the investigator's representative, I have expl<br>the procedures, the possible benefits, and the risks of this Research<br>the study; and how the participant's protected health information<br>with others: | ch Study; the alternative to being in |
|---|---|
| Signature of Person Obtaining Consent and Authorization | Date |
| You have been informed about this study's purpose, procedures, por<br>alternatives to being in the study; and how your protected health in<br>shared with others. You have received a copy of this form. You have<br>questions before you sign, and you have been told that you can ask | nformation will be collected, used and e been given the opportunity to ask |
| You voluntarily agree to participate in this study. You hereby autho your protected health information as described above. By signing the your legal rights. | |
| Signature of Person Consenting and Authorizing | Date |